CLINICAL TRIAL: NCT02303496
Title: The Effects of Autologous Platelet-Rich Plasma Cream on Photoaging and Chronological Skin Aging
Brief Title: Autologous Platelet-Rich Plasma Cream for Photoaging and Chronological Skin Aging
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Ercument Ovali, Specialist, Haematology, Acibadem University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-CREAM-1
Record Dates: First submitted 2014-11-14; First posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Chronological Aging of Skin; Photoaging of Skin
Keywords: platelet rich plasma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRP Cream Application (Experimental): Application of Cream Containing Platelet Rich Plasma and Oleaginous Base
  Interventions: Biological: Platelet Rich Plasma Cream
- SW Cream Application - Placebo (Active Comparator): Application of Cream Containing Sterile Water and Oleaginous Base
  Interventions: Biological: Placebo - Sterile Water Cream

INTERVENTIONS:
Biological: Platelet Rich Plasma Cream — Cream Containing Platelet Rich Plasma and Oleaginous Base
  Arms: PRP Cream Application
Biological: Placebo - Sterile Water Cream — Cream Containing Sterile Water and Oleaginous Base
  Arms: SW Cream Application - Placebo

SUMMARY:
Human skin undergoes some morphological changes with the effects of chronological aging and photoaging, these are especially remarkable in the facial skin. Changes in pigmentation, sallowness, deep wrinkling, laxity and elastosis are the main changes seen in photoaging and chronologic aging of skin. With the increasing demand, it needs to provide new approach for the prevention and treatment of these morphological changes.

Fibroblasts have a key role on skin aging. It is known that platelet rich plasma activates the fibroblasts and increases the synthesis of collagen and other type of matrix components. Because of these specialities, platelet rich plasma is thought to be effective on skin aging.

DETAILED DESCRIPTION:
Clinical evaluation of the patients will be done for five times during 3 months. 0th day (Basal), 7th day, 15th day, 45th day and 105th day.

ELIGIBILITY:
Inclusion Criteria:

* The patient has periorbital wrinkles with Glogau Scale 3 or more

Exclusion Criteria:

* Patients with precancerous lesions
* Patients with inflammatory skin disease like rosacea, psoriasis, seborrheic eczema
* Patients with connective tissue disease like lupus erythematosus
* Patients have a cosmetic intervention to their face, like chemical peel, infrared, radio frequency, laser, fillers or botulinum toxin injections in last 6 months
* Patients who use an anti aging cream containing retinoic acid, vitamin C and peptides in last 3 months
* Pregnant or lactating females

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Global efficacy evaluations and quantitative analyzes. | T4 (105th day)
  Evaluation of deep and fine wrinkling, amount of pigmentation, amount of vascularization, clarity of skin assessment done by the patient and the investigator. Quantitative analyzes: Measurements of Antera and Cutometer.

SECONDARY OUTCOMES:
Deep and fine wrinkling, | T0 (basal condition),T1 (7th day), T2 (15th day), T3 (45th day,) T4 (105th day)
  It will be scored from 0 to 10, by patients and the investigator
Number of Participants with Adverse Events and Type of Adverse Effects. | T1 (7th day), T2 (15th day), T3 (45th day,) T4 (105th day)
  Clinical evaluation of erythema, edema, xerosis, scaling. Each item will be scored from 0 to 3 by investigator
Smell and texture of cream | T4 (105th day)
  Patient satisfaction about smell and texture of cream. Each item will be scored from 0 to 3. (0: Very Bad, 1: Bad, 2: Good, 3: Very good)
Changes from baseline and placebo group. | T0 (basal condition),T1 (7th day), T2 (15th day), T3 (45th day,) T4 (105th day)
  The percentage of change of the evaluated parameters (listed as 1-4), from baseline (T0 vs T1,T2,T3,T4) and differences from the placebo group.
Amount of pigmentation | T0 (basal condition),T1 (7th day), T2 (15th day), T3 (45th day,) T4 (105th day)
  It will be scored from 0 to 10, by patients and the investigator
Amount of vascularization | T0 (basal condition),T1 (7th day), T2 (15th day), T3 (45th day,) T4 (105th day)
  It will be scored from 0 to 10, by patients and the investigator
Clarity of skin | T0 (basal condition),T1 (7th day), T2 (15th day), T3 (45th day,) T4 (105th day)
  It will be scored from 0 to 10, by patients and the investigator

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acibadem Labcell, Istanbul, Fahrettin Kerim Gokay Saint No:49
  - Acibadem Kozyatagi Hospital, Istanbul, Inonu Saint No.20 Kozyatagi